CLINICAL TRIAL: NCT05961605
Title: Retrospective Clinical Study of COVID-19 Associated With the Condition and Treatment of Patients With Chinese Psoriasis
Brief Title: COVID-19 Associated With Psoriasis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gang Wang, MD (Other)
Responsible Party: Sponsor-Investigator, Gang Wang, MD, Chief Director of Department of Dermatology, Xijing Hospital
Organization: Xijing Hospital (Other)
Other Study IDs: XJPF202303-PSO&COVID-19
Record Dates: First submitted 2023-07-25; First posted 2023-07-27 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Psoriasis Patients; COVID-19
Keywords: psoriasis; covid-19
MeSH Terms: conditions — COVID-19; Psoriasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A retrospective analysis based on database was conducted to evaluate the correlation between covid-19 infection and the condition and treatment of psoriasis patients.

DETAILED DESCRIPTION:
Based on the patients registered in the psoriasis patient database of each center, the patients were followed up by telephone, and the severity of covid-19 infection, the change of psoriasis condition and the adjustment of treatment methods of psoriasis patients were collected for retrospective analysis.

ELIGIBILITY:
Inclusion criteria ----

1. No age limit, both male and female are accepted;
2. Psoriasis patients registered in the database;
3. Patients or their families can cooperate to complete the follow-up information survey (questionnaire, telephone, etc.) independently, and ensure the authenticity of the data provided.

Exclusion criteria ----

Patients are thought having conditions which are not appropriated for attending this clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Psoriasis patients registered in the database from January 2018 to November 2022
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
The recurrence/exacerbation of psoriasis following SARS-CoV-2 infection | March 15,2023 to May 30,2023
  The impact of SARS-CoV-2 infection on psoriasis in patients receiving different baseline therapies of psoriasis.

SECONDARY OUTCOMES:
Univariate and multivariate analyses identify risk factors with psoriasis exacerbation/recurrence after SARS-CoV-2 infection | March 15,2023 to May 30,2023
  Univariate and multivariate analyses identify risk factors with psoriasis exacerbation/recurrence after SARS-CoV-2 infection

CONTACTS AND LOCATIONS:
Overall Officials: GANG WANG, M.D., Principal Investigator — Xijing Hospital, The Fourth Military Medical University
Locations (12):
- China (12):
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Dermatology Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second Hospital of Jilin University, Changchun, Jilin
  - Dalian Dermatosis Hospital, Dalian, Liaoning
  - Xining First People's Hospital, Xining, Qinghai
  - Xijing Hospital, The Fourth Military Medical University, Xi'an, Shaanxi
  - Shanghai Skin Disease Hospital, Tongji University School of Medicine, Shanghai, Shanghai Municipality
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen, Shenzhen
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Academy of Traditional Chinese Medicine Affiliated Hospital, Tianjin, Tianjin Municipality
  - People's Hospital of Xinjiang Uygur Autonomous Region，Xinjiang Key Laboratory of Dermatology Research, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu Y, Xu Z, Zhou J, Chen A, Zhang J, Kang X, Jiang X, Lyu C, Shi C, Shi Y, Liu X, Li F, Yang B, Huang Y, Yu C, Wang G. Clinical characteristics and outcomes of psoriasis patients with COVID-19: A retrospective, multicenter cohort study in China. Chin Med J (Engl). 2024 Jul 20;137(14):1736-1743. doi: 10.1097/CM9.0000000000003024. Epub 2024 May 6. PMID 38710539